CLINICAL TRIAL: NCT02818959
Title: First in Man Study of the JenaValve TAVI Plus System Transfemoral
Acronym: CP-0001
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to inability to recruit sufficient sample size in reasonable time frame.
Sponsor: JenaValve Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JV04FIM
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases
Keywords: Aortic Valve Disease; Aortic Valve Replacement; Transcatheter; Transfemoral; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcatheter Aortic Valve Replacement (Experimental): In this study, transcatheter aortic valve replacement (TAVR) will be performed using the JenaValve Pericardial TAVR System, which is intended for use in subjects with severe aortic stenosis. The JenaValve replacement valve is placed inside the aortic valve by using a delivery system.
  Interventions: Device: JenaValve Pericardial TAVR System

INTERVENTIONS:
Device: JenaValve Pericardial TAVR System — The JenaValve Pericardial TAVI system is intended for use in subjects with symptomatic severe aortic stenosis who are at high risk for surgical aortic valve replacement.

SUMMARY:
The objective of this study is to evaluate feasibility, safety and effectiveness of the first generation transfemoral JenaValve Pericardial TAVR System (formerly named JenaValve TAVI Plus System- Transfemoral) in an elderly patient population with severe aortic stenosis who are at high risk for surgical aortic valve replacement.

DETAILED DESCRIPTION:
The study is designed as a prospective, multi-center trial conducted at 2 centers in Germany enrolling up to 12 subjects. Each patient will be followed for 2 years. The last patient's follow-up will end in February 2016. It is planned that the study will end in June 2016. Study endpoints are defined in accordance with the "Standardized endpoint definitions for transcatheter aortic valve implantation clinical trials: a consensus report from the Valve Academic Research Consortium (VARC-2)". These endpoint definitions combine the expertise of surgeons, interventionalists, medical cardiologists, clinical trial and other specialists and allow for comparison of different trials concerning effectiveness and safety in TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe native aortic valve stenosis
* NYHA functional class II or higher
* Increased risk for surgical aortic valve replacement
* Comply with post-operative follow-up visits and requirements

Exclusion Criteria:

* Combined aortic valve disease with severe aortic insufficiency
* Presence of moderate mitral insufficiency or previous mitral prosthesis
* Severe pulmonary hypertension
* Congenital uni- or bicuspid aortic valve
* Endocarditis or active infection
* Life expectancy < 12 months
* Need for emergency surgery for any reason

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 30 days
  30-day mortality of procedure is defined as all deaths within 30 days after implantation of the JenaValve Plus Prosthesis irrespective of the underlying cause of death.

SECONDARY OUTCOMES:
Incidence rate and standard deviation of VARC-2 Individual Safety Endpoints | Index Procedure and Immediate Post-operative
  * Myocardial Infarction
  * Stroke
  * Major Bleeding
  * Acute Kidney Injury
  * Vascular Complications
  * Conduction Disturbances and Arrhythmias
  * TAVR-related Complications

OTHER OUTCOMES:
Device Success | Index Procedure and Immediate Post-operative
  Absence of procedural mortality AND Correct positioning of a single prosthetic heart valve into the proper anatomical location AND Intended performance of the prosthetic heart valve
Clinical Outcomes through 2-year follow-up - Hemodynamic Performance | Prior to discharge, at 3, 6, 12 and 24 months
  Improvement in mean gradient and effective orifice area compared to baseline and over time as assessed by Echocardiogram
Clinical Outcomes through 2-year follow-up - NYHA Functional Classification | Prior to discharge, at 3, 6, 12 and 24 months
  Number of patients with improvement over time as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Baldus, MD, Principal Investigator — University of Koln Medical Center; Hendrik Treede, MD, Principal Investigator — University of Hamburg Medical Center
Locations (2):
- Germany (2):
  - University of Koln Medical Center, Cologne
  - University of Hamburg Medical Center, Hamburg

IPD SHARING:
Plan to Share IPD: No